CLINICAL TRIAL: NCT05760248
Title: A Randomized, Double-Blind, Bilateral Comparison Study of the Safety and Efficacy of 10XB-101 in Adult Subjects With Bilateral Flank Adiposity
Brief Title: Safety and Efficacy Study of 10XB-101 in Adults With Bilateral Flank Adiposity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: 10xBio, LLC (Industry)
Collaborators: Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 210-9452-201
Record Dates: First submitted 2023-02-27; First posted 2023-03-08 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-03

CONDITIONS: Subcutaneous Fat Disorder
Keywords: Right and Left Flank Fat
MeSH Terms: interventions — Injections

STUDY DESIGN:
Intervention Model Description: Active drug 6% vs Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: 1:1 ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 10XB-101 Solution for Injection, 6.0% (Experimental): Participants receive 10XB-101 Solution for Injection, 6.0% via subcutaneous injection up to 10 mL. Injection treatment will occur once every 4 weeks for up to 6 treatments.
  Interventions: Drug: 10XB-101 Solution for Injection, 6.0%
- Placebo Solution for Injection (Placebo Comparator): Participants receive Placebo Solution for Injection, via subcutaneous injection up to 10 mL. Injection treatment will occur once every 4 weeks for up to 6 treatments.
  Interventions: Drug: Placebo Solution for Injection (no active ingredient)

INTERVENTIONS:
Drug: 10XB-101 Solution for Injection, 6.0% — The active drug (adipolytic) given as subcutaneous injection on either the right or left flank every 4 weeks for 20 weeks.
  Other Names: 10xB-101, 6%
  Arms: 10XB-101 Solution for Injection, 6.0%
Drug: Placebo Solution for Injection (no active ingredient) — Placebo given as subcutaneous injection on either the right or left flank every 4 weeks for 20 weeks.
  Other Names: Vehicle solution
  Arms: Placebo Solution for Injection

SUMMARY:
The goal of this clinical trial is to test the safety and effectiveness of an injection study drug in decreasing bilateral flank adiposity.

The main question it aims to answer is:

•How safe and effective is the injection study drug in removing bilateral flank adiposity compared to a placebo?

Participants will be:

* Be given injections every month for 5 months over the right and left flanks.
* Be asked to be seen in the clinic for 13 visits and 3 phone call visits during a duration of 1 year.

DETAILED DESCRIPTION:
Fifteen subjects with bilateral flank adiposity will be enrolled across 1-3 sites in the USA.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or non-pregnant female 18 to 55 years old.
* Subject has provided written informed consent.
* Subject has qualifying fat evaluation and skin laxity scores on each right and left flanks.
* Subject has had a stable body weight for the past 6 months prior to starting study.
* Subject is willing to undergo test article injections as directed, comply with study instructions, and commit to all follow-up visits for the duration of the study.

Exclusion Criteria:

* Subject is pregnant, lactating, or is planning to become pregnant during the study.
* Subject has loose skin in the right and left flank areas, unrepaired abdominal injury or defect, scars, tattoos, or other features that may interfere with evaluation of localized fat, in the opinion of the investigator.
* Subject has any medical condition or taking medications that affects clotting and/or platelet function
* Subject has a history of allergy or sensitivity to polidocanol or any of the other ingredients in the test articles.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-22 (Actual)

PRIMARY OUTCOMES:
Volumetric measurements | 24 weeks after final injection treatment
  Change from Baseline until end of study. Volumetric measurements will be obtained on each right and left flanks thru a standard photographic assessment.
Flank Skin Laxity Scale (FSLS) | 24 weeks after final injection treatment
  Change from Baseline on each flank after final treatment. Flank Skin Laxity Scale (FSLS) is a 4 point scale, with a score of 0 for no skin folds, and a score of 3 for severe or worse skin folds.A higher score means a worse outcome.
Clinician Global Impression of Change (CGIC) | 24 weeks after final injection treatment
  Change from Baseline on each flank after final treatment. Clinician Global Impression of Change (CGIC) is a 7-point bi-directional scale with 1 as much improved and 7 as much worse.
Patient Global Impression of Change (PGIC) | 24 weeks after final injection treatment
  Change from Baseline on each flank after final treatment. Patient Global Impression of Change (PGIC) is a 7-point bi-directional scale with 1 as much improved and 7 as much worse.

CONTACTS AND LOCATIONS:
Overall Officials: John Dobak, M.D., Study Chair — 10xBio, LLC
Locations (2):
- United States (2):
  - Site #01, Rolling Meadows, Illinois
  - Site #02, New Brighton, Minnesota

IPD SHARING:
Plan to Share IPD: No